CLINICAL TRIAL: NCT02456922
Title: A Performance Evaluation of the Harmony 1 Sensors in Adults and Pediatrics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: For administraive reasons
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CEP301
Record Dates: First submitted 2015-05-12; First posted 2015-05-29 (Estimated); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Type 1 Diabetes; Type 2 Diabetes; Harmony 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Group A (Other): Subjects wearing Harmony 1 Sensor for up to 10 days.
  Interventions: Device: Harmony 1 Sensor

INTERVENTIONS:
Device: Harmony 1 Sensor — Use of Harmony 1 Sensor over 10 days in arm and abdomen and used with the Guardian Mobile App in subjects aged 2-75 years who have had a diagnosis of type 1 or type 2 diabetes for at least one year.

SUMMARY:
The purpose of this study is to demonstrate the performance of the Harmony 1 Sensor in subjects age 2 - 75 years

DETAILED DESCRIPTION:
This study is a multi-center, randomized, prospective single-sample correlational design without controls. A total of up to 310 previously-diagnosed type 1 or 2 diabetes subjects will be enrolled in order to have 160 subjects complete frequent sample testing at up to 17 centers. Subjects will wear Harmony 1 sensors used with the Guardian Mobile application.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 2-75 years of age at time of screening
* A clinical diagnosis of type 1 or 2 diabetes for a minimum of 12 months duration as determined via medical record or source documentation by an individual qualified to make a medical diagnosis
* Adequate venous access as assessed by investigator or appropriate staff
* Subjects participating in the high and low glucose challenges must have an established insulin carbohydrate ratio(s) and insulin sensitivity ratio. (The term "established" refers to a ratio that has been previously defined and tested prior to screening visit). Subjects without established ratios may participate under observation only.

Exclusion Criteria:

* Subject will not tolerate tape adhesive in the area of Harmony 1 Sensor placement as assessed by qualified individuals
* Subject has any unresolved adverse skin condition in the area of Harmony 1 Sensor or device placement (e.g., psoriasis, rash, Staphylococcus infection)
* Subject is actively participating in an investigational study (drug or device) wherein they have received treatment from an investigational study (drug or device) in the last 2 weeks
* Subject is female and has a positive pregnancy screening test
* Females of child bearing age and who are sexually active should be excluded if they are not using a form of contraception deemed reliable by investigator
* Subject is female and plans to become pregnant during the course of the study
* Subject has had a hypoglycemic seizure within the past 6 months
* Subject has had hypoglycemia resulting in loss of consciousness within the past 6 months prior to screening visit
* Subject has had an episode of diabetic ketoacidosis (DKA) within the past 6 months prior to screening visit.
* Subject has a history of a seizure disorder
* Subject has central nervous system or cardiac disorder resulting in syncope
* Subject has a history of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack (TIA), cerebrovascular accident (CVA), angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
* Subject has a hematocrit (Hct) lower than the normal reference range
* Subject has a history of adrenal insufficiency

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Harmony 1 Sensor accuracy | 10 days
  Sensor accuracy will be evaluated compared to YSI plasma glucose values during frequent sample testing. A within 30% mean agreement rate (±22.5 mg/dL when Reference BG ≤ 75 mg/dL) between sensor and YSI will be evaluated against the null Hypothesis for varying glucose ranges.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Brazg, MD, Principal Investigator — Rainier Clinical Research Center; Mark Christiansen, MD, Principal Investigator — Diablo Clinical Research; Timothy Bailey, MD, Principal Investigator — AMCR Institute; Satish Garg, MD, Principal Investigator — Barbara Davis Center; Robert Slover, MD, Principal Investigator — Barbara Davis Center; Kevin Kaiserman, MD, Principal Investigator — SoCal Diabetes; Bruce Bode, MD, Principal Investigator — Atlanta Diabetes Associates; Luis Casaubon, MD, Principal Investigator — Texas Diabetes & Endocrinology

IPD SHARING:
Plan to Share IPD: No